CLINICAL TRIAL: NCT00244829
Title: A Multicenter Pilot Study Evaluating the Safety and Efficacy of Imatinib as Post-Transplant Therapy for High- Risk Philadelphia Chromosome-Positive Leukemias
Brief Title: Imatinib Mesylate After a Donor Stem Cell Transplant in Treating Patients With Philadelphia Chromosome-Positive Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 1867.00; FHCRC-1867.00; CDR0000355118 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: imatinib mesylate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving imatinib mesylate after a donor stem cell transplant may prevent the recurrence of Philadelphia chromosome-positive leukemia.

PURPOSE: This phase I/II trial is studying the side effects of giving imatinib mesylate after a donor stem cell transplant and to see how well it works in treating patients with Philadelphia chromosome-positive leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of adjuvant imatinib mesylate after allogeneic hematopoietic stem cell transplantation (AHSCT) in patients with high-risk Philadelphia chromosome-positive leukemia.

Secondary

* Determine the bcr/abl transcript load during the first 90 days after AHSCT in patients treated with this drug from the time of engraftment.
* Determine the 1-year survival of patients treated with this drug.

OUTLINE: This is an open-label, pilot, multicenter study.

Beginning within 14-30 days after allogeneic stem cell transplantation, patients receive oral imatinib mesylate once daily until 1 year after transplantation. Treatment continues in the absence of unacceptable toxicity or disease progression.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute lymphoblastic leukemia or chronic myeloid leukemia (CML) characterized by p^190 and/or p^210 bcr/abl gene rearrangement
  * Accelerated or blastic phase CML
  * CML in second or greater chronic phase
* No imatinib mesylate-resistant leukemia
* Planned allogeneic hematopoietic stem cell transplantation

  * Availability of an appropriately matched related or unrelated donor
  * Autologous or nonmyeloablative transplantation is not allowed
* None of the following within 4 days after the date of neutrophil engraftment*:

  * More than 5% marrow blasts
  * Circulating peripheral blood leukemic blasts
  * Aberrant antigen expression on marrow myeloblasts ≥ 1% by multidimensional flow cytometric assay
  * Presence of bcr/abl in > 5% of marrow interphase nuclei by fluorescent in situ hybridization
  * More than 1 of 20 Philadelphia chromosome-positive marrow metaphases
  * CNS involvement by leukemia NOTE: *The date of neutrophil engraftment is defined as the second consecutive day at which the peripheral blood absolute neutrophil count exceeds 500/mm3

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* At least 2 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 1,200/mm^3 (use of filgrastim [G-CSF] allowed)

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known imatinib mesylate hypersensitivity
* No other disease that severely limits life expectancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety at 90 days following transplant

SECONDARY OUTCOMES:
BCR/ABL transcript load at 90 days following transplant
Standard management of progressive minimal residual disease at 90 days following transplant
Survival at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Carpenter, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Fred Hutchinson Cancer Research Center, Seattle, Washington